CLINICAL TRIAL: NCT03750461
Title: Stoma Closure and Reinforcement (SCAR) Trial - A Single Center Pilot Study of the Safety of a Mesh Reinforcement of Ileostomy Closure to Prevent Hernia Formation in Left Sided Colon and Rectal Cancer Patients
Brief Title: Stoma Closure and Reinforcement Trial
Acronym: SCAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Hitchcock Foundation (Other)
Responsible Party: Principal Investigator, Matthew Z. Wilson, Assistant Professor of Surgery, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: D18101
Record Dates: First submitted 2018-11-13; First posted 2018-11-23 (Actual); Results first posted 2022-03-10 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Colon Cancer; Rectal Cancer; Ileostomy - Stoma
Keywords: ileostomy; hernia; rectal cancer; colon cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Hernia

STUDY DESIGN:
Intervention Model Description: Modified Simon-Two Step. An initial cohort of 5 patients will be enrolled and treated sequentially with 30 day follow-up. If stopping criteria are not met, the cohort will be expanded to an additional 15 patients followed concurrently for the duration of the study period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention (Experimental): Patients undergoing mesh implantation during ileostomy closure to reinforce the abdominal wall
  Interventions: Device: Mesh Implantation

INTERVENTIONS:
Device: Mesh Implantation — Implantation of permanent mesh (BARD Soft Mesh) into the abdominal wall for reinforcement to prevent hernia formation

SUMMARY:
Hernia formation at sites of ostomy closure is a common complication. The investigator believes that using evidence based hernia repair techniques as a preventive measure during closure of ostomies will reduce the incidence of hernia formation. In this trial, the investigator will pilot a novel technique of large pore monofilament polypropylene mesh reinforcement of the abdominal wall defects that remain after closure of an ileostomy to evaluate for safety and begin to evaluate the effectiveness compared to standard techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18years
2. Patient is undergoing closure of loop ileostomy
3. Patient has a diagnosis of left sided colon or rectal cancer treated with resection and diverting loop ileostomy
4. Patient has been evaluated by a qualified surgeon and found to be a suitable candidate for surgery

Exclusion Criteria:

1. Pre-existing systemic infection at the time of ileostomy takedown
2. Cirrhosis, chronic renal failure requiring dialysis, or collagen disorder
3. On current immunosuppression (anti-tumor necrosis factor (TNF) agents, chemotherapy, or prednisone >10mg/day)
4. Previous abdominal hernia repair with mesh placement
5. Concurrent procedures in addition to closure of diverting loop ileostomy
6. Ileostomy closure not completed through the previous stoma site (i.e. those requiring exploratory laparotomy for closure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Z Wilson, MD, Msc, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients (Interventional group)with left sided CRC who underwent proximal diversion with a LI as part of their surgical therapy were recruited from the clinical practice of the Division of Colon and Rectal Surgery at DHMC between January 2019 and November 2020.
  Historical Controls were patients diagnosed with colorectal cancer and who underwent stoma reversals from January 1, 2011, to December 31, 2018 from the clinical practice of the Division of Colon and Rectal Surgery at DHMC.
Pre-assignment Details: 24 Adult patients with left-sided colon and rectal cancer treated with resection and diverting loop ileostomy were eligible to participate. 4 participants declined participation and were not enrolled.
  Historical Controls. Data for only those who met the inclusion criteria was collected. Data collected was only relevant to the Primary endpoint, and additional follow-up date was no collected beyond the data needed for analysis for the primary outcome measure.
Groups:
- Historical Controls: Patients diagnosed with colon or rectal cancer, identified by relevant International Classification of Disease 9/10 codes, and who underwent a stoma reversal procedure, identified by pertinent current procedural terminology (CPT) codes.
Period: Overall Study
Arm/Group | Intervention | Historical Controls
Started | 20 | 92
Primary Endpoint | 20 | 92 (Considered study completion for the Historical Controls.)
Secondary Endpoint | 19 | 0 (Not applicable for the historical controls.)
Completed (Ongoing Follow-up) | 19 | 0 (Not applicable for the historical controls; no follow-up data was collected.)
Not Completed | 1 | 92

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Historical Controls | Total
Number analyzed (Participants) | 20 | 92 | 112
Age, Continuous [Mean (Full Range); unit: years] | 62 [47 to 85] | 58 [27 to 92] | 60 [27 to 92]
Age, Customized [Number; unit: years]
  Mean | 62 | 58 | 120
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 81 | 89
  Male | 12 | 11 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 19 | 91 | 110
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 92 | 112
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.19 (7.9) | 27.3 (4.95) | 28.245 (6.425)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Wound Occurrences
Description: Incidence of wound occurrences (defined as superficial surgical site infection [s-SSI], deep surgical site infection [d-SSI], organ space surgical site infection [O-SSI], dehiscence, and seroma formation) at 30 days, with particular attention to wound occurrences requiring procedural intervention, including but not limited to, operative debridement, radiographically guided drain placement, or excision of the mesh will be assessed.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 20
Participants | 0

2. Primary Outcome: Number of Participants With Wound Occurrences in Current Study Compared to Historical Controls
Description: The incidence of wound occurrences (defined as superficial surgical site infection [s-SSI], deep surgical site infection [d-SSI], organ space surgical site infection [O-SSI], dehiscence, and seroma formation) at 30days, with particular attention to wound occurrences requiring procedural intervention, including but not limited to, operative debridement, radiographically guided drain placement, or excision of the mesh will be compared to historical controls.
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Intervention | Historical Controls
Number analyzed (Participants) | 20 | 92
participants
  superficial wound infection | 0 | 5
  deep wound infection | 0 | 0
  organ/space infection | 0 | 4
  wound disruption | 0 | 0

3. Secondary Outcome: Preliminary Efficacy Based on Number of Participants With Hernia Formation
Description: Evaluation of the incidence of hernia formation at the ileostomy site on a prospective basis at 30 days and 6 month intervals thereafter until two years from the date of ileostomy closure using computed tomography and clinical examination.
Time Frame: 30 days, and then 6 months post procedure
Population: One participant was lost to follow-up due to declining cancer surveillance.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 20
Participants
  30 Days post procedure | 0
  6 months post procedure: number analyzed (Participants) | 19
  6 months post procedure | 0

4. Secondary Outcome: Bowel Function After Mesh Implantation
Description: Patient will be evaluated with regards to their bowel function outcomes utilizing the Colorectal Function Outcome (COREFO) instrument to evaluate bowel function. Score range is 0-100, Higher score indicates worse bowel function.
Time Frame: 2 years
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 20
units on a scale | 12 [10 to 30]

5. Secondary Outcome: Quality of Life After Mesh Implantation
Description: Patient will be evaluated with regards to their quality of life outcomes utilizing the Promis SF 2.0 8a Ability to Participate in Social Roles and Activities instrument. Score range is 0-40, Higher scores represents better quality of life
Time Frame: 2 years
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 20
units on a scale | 33 [15 to 40]

ADVERSE EVENTS:
Time Frame: From date of surgery to follow-up at approximately 2 years.
Description: Interventional arm: Adverse events were collected for surgical site occurrences (surgical site infection, mesh infection, delayed wound healing), fascial dehiscence, seroma, hematoma, cellulitis or enterocutaneous fistula, or return to the operating room for mesh removal.
  Historical Controls: Only adverse events relating to wound or organ/space infection and wound disruption were collected.
Arm/Group | Intervention | Historical Controls
All-Cause Mortality (participants affected / at risk) | 1/20 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/92
Other Adverse Events (participants affected / at risk) | 2/20 | 9/92
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=20) | Historical Controls (N=92)
Ogilvie's syndrome (Gastrointestinal disorders) | 1 (1) | 0
Myocardial infarction (Cardiac disorders) | 1 (1) | 0
superficial wound infection (Infections and infestations) | 0 | 5 (5)
organ/space infection (Infections and infestations) | 0 | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-09): https://cdn.clinicaltrials.gov/large-docs/61/NCT03750461/Prot_SAP_000.pdf